CLINICAL TRIAL: NCT02924350
Title: A Clinical Study Investigating the Efficacy of an Occluding Dentifrice in Providing Relief From Dentinal Hypersensitivity
Brief Title: The Efficacy of an Occluding Dentifrice in Providing Relief From Dentinal Hypersensitivity (DH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 207212
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-02

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Tin Fluorides; fluorophosphate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test dentifrice containing stannous fluoride (Experimental): All the participants in the test arm applied test dentifrice on their two test teeth using their finger, followed by brushing these test teeth, followed by brushing the whole mouth using test dentifrice. Participants brushed their teeth for 3 days twice daily (morning /evening).
  Interventions: Other: Stannous fluoride
- Control dentifrice containing sodium monofluorophosphate (Active Comparator): All the participants in the control arm applied control dentifrice on their two test teeth using their finger, followed by brushing these test teeth, followed by brushing the whole mouth using control dentifrice. Participants brushed their teeth for 3 days twice daily (morning /evening).
  Interventions: Other: Sodium monofluorophosphate

INTERVENTIONS:
Other: Stannous fluoride — Supervised direct application (Day 0): Participants applied a pea-sized dose of test dentifrice to each of the 2 qualifying test teeth using their washed and clean finger to gently rub the dentifrice into the tooth's cervical margin for 60 sec. No rinsing was permitted after treatment.
  Supervised brushing (Day 0, before leaving the site) and Home use (3 days): after dosing a dry toothbrush with a full strip of dentifrice, participants brushed each of the 2 qualifying test teeth first, followed by their whole mouth for at least 60 sec. Participants were permitted to rinse with 5 mL tap water (room temperature) for 5 sec. maximum after brushing on supervised brushing (Day 0) and were also permitted to rinse with tap water after brushing on home use (3 days).
  Arms: Test dentifrice containing stannous fluoride
Other: Sodium monofluorophosphate — Supervised direct application (Day 0): participants applied a pea-sized dose of control dentifrice to each of the 2 qualifying test teeth using their washed and clean finger to gently rub the dentifrice into the tooth's cervical margin for 60 sec. No rinsing was permitted after treatment.
  Supervised brushing (Day 0, before leaving the site) and home use (3 days): after dosing a dry toothbrush with a full strip of dentifrice, participants brushed their whole mouth thoroughly for at least 60 sec. Participants were permitted to rinse with 5mL tap water (room temperature) for 5 sec. maximum after brushing in supervised brushing on Day 0 and were also permitted to rinse with tap water after brushing on home use (3 days).
  Arms: Control dentifrice containing sodium monofluorophosphate

SUMMARY:
This single center study will investigate the efficacy of an experimental stannous fluoride containing dentifrice in relieving DH compared with a standard fluoride dentifrice after short term use.

DETAILED DESCRIPTION:
This was a single centre, 3 day, randomised, examiner blind, two treatment arm, parallel design, stratified (by maximum baseline Schiff sensitivity score of the two selected test teeth), controlled study in participants with at least two sensitive teeth that met the study criteria at the Screening and Baseline visits. Study participants were in good general health, with pre-existing self-reported and clinically diagnosed tooth sensitivity at screening. Participants were assessed at Baseline (pre-treatment), immediately after first treatment, and after 3 days twice daily treatment, to monitor clinical efficacy and safety. At the Screening visit, participants gave their written informed consent to participate in the study. Demography, medical history and concomitant medications were recorded, followed by an oral examination which included an oral soft tissue (OST) examination and assessments to determine eligible teeth. Eligible participants were supplied with a regular fluoride dentifrice (containing 1450 parts per million (ppm) fluoride as sodium monofluorophosphate) to use twice daily (morning and evening) during the acclimatisation period (4-8 weeks) between Screening and Baseline. Each brushing occasion was recorded in a product use diary. First use of the acclimatisation dentifrice was carried out under supervision at the study site. At Baseline (Day 0, pre-treatment), eligibility to continue was assessed. Following an OST examination, tooth sensitivity was assessed (first to a tactile stimulus [Yeaple probe, maximum 20 grams (g) pressure], and then to an evaporative air stimulus [Schiff sensitivity scale]), and the inclusion/exclusion criteria were reviewed. Eligible participants were stratified and randomised to treatment. First use of allocated study treatment was by direct application to the 2 selected test teeth, and was carried out under supervision at the study site. The sensitivity of the 2 test teeth was reassessed immediately post-treatment, first to a tactile stimulus (Yeaple probe, maximum 80g pressure), and then to an evaporative air stimulus (Schiff sensitivity scale). Participants completed a supervised whole mouth brushing with their allocated study treatment prior to leaving the study site. Sensitivity was re-assessed after 3 days twice daily treatment. Each use of study treatment was recorded in a product use diary. Adverse events (AEs) were documented from completion of the first use of acclimatisation dentifrice until 5 days following last administration of study product. Incidents were documented from completion of the first use of investigational product until 5 days following last administration of study product.

ELIGIBILITY:
Inclusion Criteria:

* Consent: Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form
* Aged 18-65 years inclusive
* Understands and is willing, able and likely to comply with all study procedures and restrictions
* Good general and mental health with, in the opinion of the investigator or medically qualified designee: a) No clinically significant and relevant abnormalities of medical history or oral examination. b) Absence of any condition that would impact on the participants safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements
* At Visit 1 (Screening): a) Self-reported history of DH lasting more than six months but not more than 10 years. b) Minimum of 20 natural teeth. c) Minimum of 2 accessible non-adjacent teeth (incisors, canines, pre-molars), preferably in different quadrants, that meet all of the following criteria: -Signs of facial/cervical gingival recession and/or signs of erosion or abrasion (EAR). -Tooth with modified gingival index (MGI) score =0 adjacent to the test area (exposed dentine) only [Lobene, 1986] and a clinical Tooth with signs of sensitivity measured by qualifying evaporative air assessment (Y/N response) mobility of ≤1, -Tooth with signs of sensitivity measured by qualifying evaporative air assessment (Y/N response)
* At Visit 2, Baseline (Pre-treatment):Minimum of two, non-adjacent accessible teeth (incisors, canines, pre-molars), that meet all of the following criteria:-Tooth with signs of sensitivity, measured by qualifying tactile stimulus (Yeaple ≤ 20g) and evaporative air assessment (Schiff sensitivity score ≥ 2)
* Teeth which meet the EAR, MGI and mobility inclusion criteria and none of the dentition exclusion criteria at Screening should be assessed by tactile stimulus at Visit 2. Those teeth which meet the required tactile threshold (Yeaple ≤ 20g) should then be assessed by evaporative air stimulus. When two teeth that meet the study criteria are identified, no further testing is necessary

Exclusion Criteria:

* A woman who is known to be pregnant or who is intending to become pregnant over the duration of the study
* A woman who is breast-feeding
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit
* Previous participation in this study
* Participation in study 205084
* Recent history (within the last year) of alcohol or other substance abuse
* An employee of the sponsor or the study site or members of their immediate family The site for this protocol is the Clinical trials Unit in the Bristol Dental School and Hospital. Employees of the Bristol Dental School and Hospital not associated with the Clinical Trials unit are eligible to participate
* Presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes
* Any condition which, in the opinion of the investigator, causes xerostomia
* Dental prophylaxis within 4 weeks of Screening
* Tongue or lip piercing or presence of dental implants on the selected Test Teeth
* Gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of Screening, scaling or root planning within 3 months of Screening
* Vital teeth bleaching within 8 weeks of Screening
* Desensitizing treatment within 8 weeks of Screening (professional sensitivity treatments and non-dentifrice sensitivity treatments)
* Tooth with evidence of current or recent caries, or reported treatment of decay within 12 months of Screening
* Tooth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns or veneers, orthodontic bands or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine
* Sensitive tooth not expected to respond to treatment with an over-the-counter dentifrice in the opinion of the investigator
* Use of an oral care product indicated for the relief of dentine hypersensitivity within 8 weeks of screening (participants will be required to bring their current oral care products to the site in order to verify the absence of known anti-sensitivity ingredients)
* Daily doses of medication/treatments which, in the opinion of the investigator, could interfere with the perception of pain. Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilisers, anti-depressants, mood-altering and anti-inflammatory drugs
* Currently taking antibiotics or has taken antibiotics within 2 weeks of Baseline
* Daily dose of a medication which, in the opinion of the investigator, is causing xerostomia
* Any participants who, in the judgment of the investigator, should not participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bristol, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one center in the United Kingdom.
Pre-assignment Details: A total of 246 participants were screened, out of which 205 participants enrolled in the study. 41 of screened participants were not enrolled because of screening failure. Of 205 enrolled participants, 204 were randomized in study, one participant was not randomized due to lost to follow up.
Period: Overall Study
Arm/Group | Test Dentifrice Containing Stannous Fluoride | Control Dentifrice Containing Sodium Monofluorophosphate
Started | 102 | 102
Completed | 102 | 100
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Dentifrice Containing Stannous Fluoride | Control Dentifrice Containing Sodium Monofluorophosphate | Total
Number analyzed (Participants) | 102 | 102 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.8 (6.61) | 22.2 (5.12) | 22.5 (5.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 74 | 139
  Male | 37 | 28 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 5 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 85 | 90 | 175
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Schiff Sensitivity Score on Day 3
Description: The examiner indicated the participant's response to the evaporative air stimulus, after the stimulation of each individual tooth, using the Schiff Sensitivity Scale as follows: 0=Participant does not respond to air stimulation, 1=Participant responds to air stimulus but does not request discontinuation of stimulus, 2=Participant responds to air stimulus and requests discontinuation or moves from stimulus, 3=Participant responds to stimulus, considers stimulus to be painful and requests discontinuation of the stimulus. A reduction in Schiff Sensitivity score indicates improvement in sensitivity.
Time Frame: Baseline, Day 3
Population: Intent to treat (ITT) population, defined as all participants who were randomized, received study treatment at least once & provided at least one post-baseline (post treatment) assessment of efficacy. Number of participants analyzed is from ITT population evaluated at specific time points for each treatment arms respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Dentifrice Containing Stannous Fluoride | Control Dentifrice Containing Sodium Monofluorophosphate
Number analyzed (Participants) | 102 | 100
score on a scale | -1.37 (0.520) | -0.45 (0.443)
Statistical Analysis 1: Comparison: Test Dentifrice Containing Stannous Fluoride vs Control Dentifrice Containing Sodium Monofluorophosphate; Test type: Other; p < .0001, ANCOVA; ANCOVA: change from baseline in Schiff sensitivity score as response and treatment as a factor and baseline Schiff sensitivity score as a covariate; Least square (LS) mean difference = -0.924, 95% CI 2-sided [-1.0547 to -0.7927] — Difference is first named dentifrice minus second named dentifrice such that a negative difference favors first named dentifrice

2. Secondary Outcome: Change From Baseline (Day 0 Pre-treatment) in Schiff Sensitivity Score on Day 0 (After 60 Seconds of Single Direct Application)
Description: as for outcome 1
Time Frame: At Baseline (Day 0 pre-treatment) and after 60 seconds of single direct application on Day 0
Population: ITT population, defined as all participants who were randomized, received study treatment at least once & provided at least one post-baseline(post treatment) assessment of efficacy. Number of participants analyzed is the ITT population evaluated at specific time points for each treatment arms respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Dentifrice Containing Stannous Fluoride | Control Dentifrice Containing Sodium Monofluorophosphate
Number analyzed (Participants) | 102 | 102
score on a scale | -0.63 (0.536) | -0.38 (0.413)

3. Secondary Outcome: Change From Baseline (Day 0 Pre-treatment) in Tactile Threshold on Day 0 (After 60 Seconds of Single Direct Application) and Day 3
Description: The examiner assessed the response to tactile sensitivity using a Yeaple probe which allowed the application of a known force to the dentin surface, starting at 10gram (g) and raised in increments of 10g until the tactile threshold or maximum force was reached. The tactile threshold for each tooth was determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gave two consecutive 'yes' responses were recorded as the tactile threshold. Higher tactile threshold means less sensitive tooth. At baseline, the maximum force used was 20g; at all subsequent visits, it was 80g.
Time Frame: At Baseline (Day 0 pre-treatment), after 60 seconds of single direct application on Day 0 and Day 3
Population: ITT population, defined as all participants who were randomized, received the study treatment at least once and provided at least one post-baseline (post treatment) assessment of efficacy. Number of participants analyzed is from ITT population evaluated at specific time points for each treatment arms respectively.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Test Dentifrice Containing Stannous Fluoride | Control Dentifrice Containing Sodium Monofluorophosphate
Number analyzed (Participants) | 102 | 102
g
  Change from baseline on Day 0 | 15.10 (14.229) | 8.14 (9.823)
  Change from baseline on Day 3: number analyzed (Participants) | 102 | 100
  Change from baseline on Day 3 | 32.79 (17.257) | 10.45 (11.149)

ADVERSE EVENTS:
Time Frame: up to 64 days (from completion of the first use of acclimatisation dentifrice until 5 days following last administration of study product on Visit 3)
Description: The time frame for adverse event (AE) reporting was calculated as 64 days including maximum (max.) 56 days of acclimatization period (minimum 28 days and max of 56 days of regular fluoride dentifrice use in acclimatization period, in between of screening and baseline visit), followed by 3 study days and 5 follow up days.
Arm/Group | Test Dentifrice Containing Stannous Fluoride | Control Dentifrice Containing Sodium Monofluorophosphate
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/102
Other Adverse Events (participants affected / at risk) | 9/102 | 11/102
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Dentifrice Containing Stannous Fluoride (N=102) | Control Dentifrice Containing Sodium Monofluorophosphate (N=102)
Headache (Nervous system disorders) | 2 (2) | 6 (6)
Dizzines (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Seasonal Allergy (Immune system disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-08-28): https://cdn.clinicaltrials.gov/large-docs/50/NCT02924350/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT02924350/SAP_001.pdf